CLINICAL TRIAL: NCT02423239
Title: A Phase 1b Study to Assess the Safety and Anti-tumour Activity of Dexanabinol Monotherapy and Dexanabinol in Combination With Chemotherapy in Patients With Advanced Tumours
Brief Title: A Study of Dexanabinol in Combination With Chemotherapy in Patients With Advanced Tumours
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: e-Therapeutics PLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETS2101-004
Record Dates: First submitted 2015-04-09; First posted 2015-04-22 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Hepatocellular Carcinoma; Pancreatic Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Pancreatic Neoplasms | interventions — HU 211; Sorafenib; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Relapsed or refractory advanced tumours (Experimental): Patients with selected relapsed or refractory tumour types to receive single agent dexanabinol.
  Interventions: Drug: Dexanabinol
- Newly diagnosed hepatocellular carcinoma (Experimental): Patients with hepatocellular carcinoma to receive dexanabinol in combination with standard chemotherapy.
  Interventions: Drug: Dexanabinol; Drug: Sorafenib
- Newly diagnosed pancreatic cancer (Experimental): Patients with pancreatic cancer to receive dexanabinol in combination with standard chemotherapy
  Interventions: Drug: Dexanabinol; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Dexanabinol — Patients will receive dexanabinol given once a week, as a slow intravenous infusion (i.v.) over a 3 hour period
  Other Names: ETS2101; HU-211
Drug: Sorafenib — Patients will receive Sorafenib at a dose of 400 mg bid (oral administration)
  Arms: Newly diagnosed hepatocellular carcinoma
Drug: Nab-paclitaxel — Patients will receive Nab-paclitaxel at a dose of 125mg/m2 intravenous infusion
  Arms: Newly diagnosed pancreatic cancer
Drug: Gemcitabine — Patients will receive Gemcitabine at a dose of 1000mg/m2 intravenous infusion
  Arms: Newly diagnosed pancreatic cancer

SUMMARY:
This study is a trial of dexanabinol in patients with advanced tumours. The purposes of the protocol are to study different doses of the study drug to determine the maximum safe dose of the drug given in combination with standard chemotherapies and to further understand the safety of the study drug and to measure any reduction in size of patients' cancer tumour(s).

Dexanabinol is a synthetic cannabinoid which has previously undergone clinical trials for traumatic brain injury (TBI) and in subjects undergoing coronary artery bypass surgery. Currently dexanabinol is under investigation for potential anti-tumour activity in patients with advanced tumours.

ELIGIBILITY:
Inclusion Criteria

1. (i) Parts 1 and 2b (dexanabinol combination): Patients with selected histologically, cytologically or radiologically confirmed tumours that are advanced, metastatic and/or progressive, and eligible for 1st line chemotherapy.

   * HCC only: patient with Child-Pugh A stage.
   * Pancreatic cancer only: patients diagnosed with adenocarcinoma (i.e. pancreatic cancer patients with islet cell neuroplasms are excluded).

   (ii) Part 2a (dexanabinol monotherapy): Patients with histologically, cytologically or radioloigically confirmed tumours that are advanced, metastatic and/or progressive, for whom there is no effective standard therapy available.
   * Pancreatic cancer only: patients diagnosed with adenocarinoma (i.e. pancreatic cancer patients with islet cell neuroplasms are excluded).
2. Adults patients defined by age ≥ 18 years.
3. Eastern Collaborative Oncology Group (ECOG) Performance Status (PS) or 0 or 1.
4. Any acute or chronic adverse effects of prior chemotherapy or radiotherapy have resolved to < Grade 2 as determined by CTCAE v4.03 criteria, with the exception of alopecia.
5. (i) Parts 1 and 2b: Measureable disease assessed by appropriate method for each tumour type e.g. RECIST 1.1 (Eisenhauer, et al. 2009).

   (ii) Part 2a: Evaluable disease, either measureable on imaging, or with informative tumour marker(s).
6. Laboratory values at Screening:

   * Absolute neutrophil count ≥ 1.5 x 109L;
   * Platelets ≥ 100 x 109/L;
   * Total bilirubin; in 1st line pancreatic cancer (part 1 and 2b) ≤1.25 times the upper limit of normal (ULN); all other tumour types and settings except HCC ≤1.5 times ULN; in HCC ≤5 times the ULN
   * AST (SGOT) ≤2.5 times the ULN (when there is no liver tumour involvement) up to

     * 5 times the ULN (in patients with liver tumour involvement);
   * ALT (SGPT) ≤2.5 times the ULN (when there is no liver tumour involvement) up to

     * 5 times the ULN (in patients with liver tumour involvement);
   * Estimated GFR of >50 mL/min (based on the Wright formula (Wright, et al. 2001 ); and
   * Negative hCG test in women of childbearing potential
7. Have a life expectancy of >3 months.
8. Ability to give written, informed consent prior to any study-specific Screening procedures, with the understanding that the consent may be withdrawn by the patient at any time without prejudice.
9. Be willing and able to comply with the study protocol procedures.

Exclusion Criteria

1. Patient is pregnant or breast feeding.
2. History of clinically significant cardiac condition, including ischemic cardiac event, myocardial infarction or unstable cardiac disease within 3 months of Cycle 1, Day 1.
3. Known brain metastases.
4. (i) Parts 1 and 2b (dexanabinol combination): Prior systemic chemotherapy.

   (ii) Part 2a (dexanabinol monotherapy): Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to Cycle 1, Day 1 for solid tumours (with the exception of hydroxyurea, which must be discontinued at least 24 hours prior to Cycle 1, Day 1). Localised palliative radiotherapy is permitted for symptom control.
5. Major surgery within 4 weeks prior to Cycle 1, Day 1; bone marrow transplant within 100 days prior to Cycle 1, Day 1.
6. Known human immunodeficiency virus positivity.
7. Active hepatitis B or C or other active liver disease (other than malignancy) (applies to all tumours types enrolled except HCC).
8. Use of any investigational agents within 4 weeks of Cycle 1, Day 1.
9. Any active, clinically significant, viral, bacterial, or systemic fungal infection within 4 weeks prior to Cycle 1, Day 1.
10. History of significant chronic or recurrent infections requiring treatment or any uncontrolled intercurrent illness that would jeopardize patient safety, interfere with the objectives of the protocol, or limit patient compliance with study requirements, as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of dexanabinol given in combination with standard chemotherapies | For 29 days from the day of first dose
  Patients will be sequentially assigned to increasing doses of dexanabinol to establish the MTD (or maximum administered dose (MAD)). 3 patients will be enrolled to a cohort to assess each dose level. Dose escalation to a cohort of 3 new patients will occur when all patients in the previous cohort have completed the first cycle i.e. the first four doses followed by observation through to day 29 and no dose limiting toxicity (DLT) has occurred.
Number of adverse events (AEs) in patients receiving dexanabinol monotherapy | From start of dosing until 30 days ± 3 days post last dose of dexanbinol
  AEs will be graded according to the NCI CTCAE v4.03 for cancer clinical trials.
Number of adverse events (AEs) in patients receiving dexanabinol in combination with standard chemotherapies | From start of dosing until 30 days ± 3 days post last dose of IMP
  AEs will be graded according to the NCI CTCAE v4.03 for cancer clinical trials.

SECONDARY OUTCOMES:
Area under curve (AUC) of dexanabinol and (where applicable) combination chemotherapy | Cycle 1 Day 1 and Day 8 pre-dose (0h); 1, 2, 3h (i.e. immediately prior to end infusion) post start of infusion; 5, 10, 15, 30 min post-end infusion; 1, 2, 3, 4, 6, 8, 10 and 24h post-end infusion; day 15 immediately prior to and at end of IMP infusion
Maximum concentration (Cmax) of dexanabinol and (where applicable) combination chemotherapy | Cycle 1 Day 1 and Day 8 pre-dose (0h); 1, 2, 3h (i.e. immediately prior to end infusion) post start of infusion; 5, 10, 15, 30 min post-end infusion; 1, 2, 3, 4, 6, 8, 10 and 24h post-end infusion day 15 immediately prior to and at end of IMP infusion
Minimum concentration (Cmin) of dexanabinol and (where applicable) combination chemotherapy | Cycle 1 Day 1 and Day 8 pre-dose (0h); 1, 2, 3h (i.e. immediately prior to end infusion) post start of infusion; 5, 10, 15, 30 min post-end infusion; 1, 2, 3, 4, 6, 8, 10 and 24h post-end infusion day 15 immediately prior to and at end of IMP infusion
Tumour response ( RECIST 1.1, assessment by CT or MRI) | Participants will be followed until objective disease progression as per the RECIST v1.1 criteria, an expected average of four months
  Tumour response evaluation using RECIST 1.1 (assessment by CT or MRI).

CONTACTS AND LOCATIONS:
Locations (13):
- Germany (5):
  - University Hospital Bonn, Study Center Bonn (SZB) Clinical Study Core Unit Institute of Clinical Chemistry and Clinical Pharmacology University Hospital Bonn, Sigmund-Freud-Str. 25, Bonn
  - Universitätsklinikum Hamburg-Eppendorf II. Medizinischen Klinik Martinistr. 52, Hamburg
  - Klinikum der Ruhr-Universitaet Bochum, Medizinische Klinik III - Hämatologie/Onkologie Marien Hospital Herne Universitätsklinikum der Ruhr-Universität Bochum Hölkeskampring 40, Herne
  - Klinikum der Universität München, Universitätsklinikum Großhadern Medizinische Klinik und Poliklinik III AG Onkologie Marchioninistr. 15, München
  - UNIFONTIS Praxis fur Integrative Onkologie, Hoppe-Seyler-Straße 6,, Tübingen
- Poland (2):
  - Osrodek Medyczny SAMARYTANIN, ul. Kazimierza Pużaka 11, Opole
  - Wojewodzki Szpital Zespolony w Toruniu, ul. Św. Józefa 53-59, Torun
- Spain (3):
  - Hospital Universitario Virgen de la Victoria, Servicio de Oncología Médica Campus de Teatinos,, Málaga, Malaga
  - START MADRID-FJD, Hospital Fundación Jiménez Díaz, Av Reyes Católicos 2, Floor 1 28040, Madrid
  - Hospital Universitario Virgen del Rocio, Hospital Universitario Virgen del Rocío Oncología Médica Avda. Manuel Siurot,, Seville
- United Kingdom (3):
  - Beatson West of Scotland Cancer Centre, 1053 Great Western Rd,, Glasgow
  - St James's Hospital, Cancer Research UK Clinical Centre/Section of Oncology, Beckett St,, Leeds
  - Freeman Hospital, Sir Bobby Robson Cancer Trials Research Centre, Freeman Road, High Heaton,, Newcastle upon Tyne